CLINICAL TRIAL: NCT01333514
Title: Carbohydrate Consumption as a Factor in Aspart Dosing Compared to the Regularly Used Standard of Care Basis of Dosing Aspart in the Inpatient Setting (CARB)
Brief Title: Carbohydrate Consumption as a Factor in Aspart Dosing
Acronym: CARB
Status: Terminated | Phase: Phase 4 | Type: Interventional
Sponsor: Rush University Medical Center (Other)
Responsible Party: Principal Investigator, Chung Kay Koh, M.D., Rush University Medical Center
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 10040503
Record Dates: First submitted 2011-04-08; First posted 2011-04-12 (Estimated); Results first posted 2023-05-01 (Actual); Last update posted 2023-05-01 (Actual); Status verified 2023-04

CONDITIONS: Diabetes
Keywords: diabetes; prandial; insulin; aspart; carbohydrate; inpatient; novolog
MeSH Terms: conditions — Diabetes Mellitus; Insulin Resistance | interventions — Insulin Aspart

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Carbohydrate based prandial insulin dosing (Experimental): Subjects will received prandial insulin based on the amount of carbohydrates consumed.
  Interventions: Drug: aspart
- Usual Care Prandial insulin dosing (Active Comparator): Subjects will received prandial insulin if they consume 50% or more of their meal-tray as is the usual care.
  Interventions: Drug: aspart- Insulin

INTERVENTIONS:
Drug: aspart — Subjects will received aspart insulin subcutaneously based on the amount of carbohydrates consumed based on the formula 0.1 units/kg X (grams of carbohydrate eaten/75 grams carbohydrate)
  Other Names: Novolog
  Arms: Carbohydrate based prandial insulin dosing
Drug: aspart- Insulin — 0.1 units/kg of Aspart insulin will be given subcutaneously TID with meals if a subject eats 50% or more of their meal-tray
  Other Names: Novolog
  Arms: Usual Care Prandial insulin dosing

SUMMARY:
Good sugar control in postoperative hospitalized patient has been shown to improve wound healing and infection rates. However, sugar control is difficult to achieve and suboptimal use of insulin is thought to be a contributory factor. Though it is known that generally the consumption of carbohydrates alone raises the blood sugar, the usual practice of dosing meal-time insulin is based on the fraction of the total meal-tray eaten which includes proteins, fats and carbohydrates. This leads to an overestimation of insulin required for a patient who consumes a portion of mainly proteins and fats on their trays or an underestimation for those eating mainly the carbohydrates on their tray. Low sugars or high blood sugars can follow respectively.

Hypothesis: The purpose of this study is to see if dosing meal-time insulin based on grams of carbohydrates consumed will result in better sugar control compared to the usual practice of dosing meal-time insulin based on percent of total meal consumed in hospitalized patients.

DETAILED DESCRIPTION:
100 research subjects are expected to be enrolled in this study, all recruited from the Rush University Medical Center surgical (non-critical) services.

As is the usual care at Rush University Medical Center, patients who have type 2 diabetes and are on insulin and or at least two oral diabetes medications are given only insulin during their inpatient stay to control their blood sugar. It is the normal practice to use only insulin the hospital instead of pills for treating your diabetes. The use of insulin would be temporary and just during your hospital stay. When you return home, you will resume using pills.

Before the study begins, a computer system will randomly assign you a number, and those numbers belong to one of two groups. The number you have been given will determine which group you will go to. Throughout the study, you will be given a standard dose of basal insulin (Lantus). This dose will be your home dose if you are already using insulin. If you are not using insulin, you will be given a dose based on your weight.

During your stay, you will be given meal trays for breakfast, lunch, and dinner, and each of the food items belonging to your meal tray will be marked with at a certain number of carbohydrates. For example, ½ cup of cottage cheese will contain 4 grams of carbohydrates and one slice of whole wheat bread will contain 14 grams of carbohydrates and one 5 oz apple will contain 21 grams of carbohydrates. A dietician will then count the total amount of carbohydrates that you consume with each meal.

If you are assigned to the investigational arm of the study, you will be given a dose of mealtime insulin (Aspart) based on the number of carbohydrates you have consumed. If you are assigned to the control arm, you will be given your standard dose of mealtime insulin, if you eat more than 50% of your tray as is the usual practice at Rush, regardless of how much carbohydrate you eat. This dose will be your home dose if you are already using insulin or calculated based on your weight.

In either arm, if meals are not given (due to additional procedures or other reasons) the insulin dose will not be given. For both arms of the study, you will be requested not to eat any snacks containing carbohydrates. Instead you may be request for snacks that do not contain carbohydrates such string cheese which the investigators will provide.

Response to these therapies will be monitored by fingerstick glucose readings, also called point-of-care glucose. Your nurses will draw capillary blood, (less than 1 ml) via fingerstick on 4 occasions: pre-breakfast, pre-lunch, pre-dinner, and post-dinner / bedtime. These values will be sent to the study investigators, who will then adjust the amount of insulin that you are given.

In addition, your doctors will check a blood test called an A1c. This test measures the average sugar level in your blood over the last 90 days. This test is done on all patients with diabetes who are hospitalized.

ELIGIBILITY:
Inclusion Criteria:

* Adults aged > or = to 18 admitted to general surgical floors, excluding the ICU, at Rush University Medical Center, regardless of race, ethnicity, gender
* Clinical diagnoses of type 2 diabetes for more than 6 months prior to admission
* Treated with insulin and/or 2 or more oral diabetic agents
* Estimated length of stay 3 days or more
* Postoperative point of care blood glucose of > 180 mg/dL

Exclusion Criteria:

* Glomerular Filtration Rate < 60 based on MDRD equation
* Pregnant patients
* Receiving parenteral or enteral nutrition
* Patients with an admitting diagnosis of hypoglycemia
* Outpatient insulin < 0.5 units/kg/day
* Inability to give consent
* Severe liver disease
* Known hypopituitarism or adrenal insufficiency
* Treatment with Prednisone at dose > 5 mg daily or its equivalent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 14 (Actual)
Dates: Start 2011-04; Primary Completion 2012-12 (Actual); Study Completion 2012-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Chung-Kay Koh, MD, Principal Investigator — Rush University Medical Center
Locations (1):
- Rush University Medical Center, Chicago, Illinois, United States

REFERENCES:
- [Background] Shilling AM, Raphael J. Diabetes, hyperglycemia, and infections. Best Pract Res Clin Anaesthesiol. 2008 Sep;22(3):519-35. doi: 10.1016/j.bpa.2008.06.005. PMID 18831301
- [Result] Cook CB, Castro JC, Schmidt RE, Gauthier SM, Whitaker MD, Roust LR, Argueta R, Hull BP, Zimmerman RS. Diabetes care in hospitalized noncritically ill patients: More evidence for clinical inertia and negative therapeutic momentum. J Hosp Med. 2007 Jul;2(4):203-11. doi: 10.1002/jhm.188. PMID 17683100
- [Result] Wexler DJ, Meigs JB, Cagliero E, Nathan DM, Grant RW. Prevalence of hyper- and hypoglycemia among inpatients with diabetes: a national survey of 44 U.S. hospitals. Diabetes Care. 2007 Feb;30(2):367-9. doi: 10.2337/dc06-1715. No abstract available. PMID 17259511
- [Result] Rabasa-Lhoret R, Garon J, Langelier H, Poisson D, Chiasson JL. Effects of meal carbohydrate content on insulin requirements in type 1 diabetic patients treated intensively with the basal-bolus (ultralente-regular) insulin regimen. Diabetes Care. 1999 May;22(5):667-73. doi: 10.2337/diacare.22.5.667. PMID 10332663
- See also: American College of Endocrinology and American Diabetes Association Consensus Statement on Inpatient Diabetes and Glycemic Control — https://linkinghub.elsevier.com/retrieve/pii/S1530891X2041818X

RESULTS

PARTICIPANT FLOW:
Groups:
- Usual Care Prandial Insulin Dosing: Subjects will received prandial insulin if they consume 50% or more of their meal-tray as is the usual care.
  aspart: 0.1 units/kg of Aspart insulin will be given subcutaneously TID with meals if a subject eats 50% or more of their meal-tray
Period: Overall Study
Arm/Group | Carbohydrate Based Prandial Insulin Dosing | Usual Care Prandial Insulin Dosing
Started | 8 | 6
Completed (One subject refused to participate after enrolling because he was not allowed to snack in between meals.) | 7 | 6
Not Completed | 1 | 0
Not completed — Withdrawal by Subject | 1 | 0

BASELINE CHARACTERISTICS:
Population: The study group had 8 subjects because due to randomization the study was selected for the next draw.
Groups:
- Total: Total of all reporting groups
Arm/Group | Carbohydrate Based Prandial Insulin Dosing | Usual Care Prandial Insulin Dosing | Total
Number analyzed (Participants) | 8 | 6 | 14
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 1 | 3 | 4
  >=65 years | 7 | 3 | 10
Age, Continuous [Mean (Standard Deviation); unit: years] | 61.5 (7.2) | 70.4 (9.4) | 66 (9.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 3 | 6
  Male | 5 | 3 | 8
Region of Enrollment [Number; unit: participants]
  United States | 8 | 6 | 14

OUTCOME MEASURES:

1. Primary Outcome: Probability of Hypoglycemia
Description: Will determine if the probability of hypoglycemia in each arm; calculation details [i.e. "Experimental Event Rate (EER) = probability of outcome occurring in experimental group = a/(a+b)"]
Time Frame: measured 4 times/day until completion of study an average of 2 days
Measure: Number; unit: probability
Arm/Group | Carbohydrate Based Prandial Insulin Dosing | Usual Care Prandial Insulin Dosing
Number analyzed (Participants) | 7 | 6
probability | 0.025 | 0.011

2. Secondary Outcome: Probability of Hyperglycemia
Description: Will determine if the probability of hyperglycemia in each arm; calculation details [i.e. "Experimental Event Rate (EER) = probability of outcome occurring in experimental group = a/(a+b)"]
Time Frame: blood sugars/4x day until completion of study, an average of 2 days
Measure: Number; unit: probability
Arm/Group | Carbohydrate Based Prandial Insulin Dosing | Usual Care Prandial Insulin Dosing
Number analyzed (Participants) | 7 | 6
probability | 0.4 | 0.329

ADVERSE EVENTS:
Time Frame: 3 months
Arm/Group | Carbohydrate Based Prandial Insulin Dosing | Usual Care Prandial Insulin Dosing
All-Cause Mortality (participants affected / at risk) | 0/7 | 0/6
Serious Adverse Events (participants affected / at risk) | 0/7 | 0/6
Other Adverse Events (participants affected / at risk) | 0/7 | 0/6

LIMITATIONS AND CAVEATS:
Early termination due to the PI becoming sick early in the study.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes